CLINICAL TRIAL: NCT00972322
Title: A Placebo-Controlled Multiple Dose Study to Evaluate the Pharmacokinetics and Pharmacokinetics of MK-8245 in Subjects With Type 2 Diabetes
Brief Title: Pharmacokinetics and Pharmacodynamics of MK-8245 in Participants With Type 2 Diabetes (MK-8245-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8245-012; MK-8245-012 (Other: Merck); 2009_655
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (5-(3-(4-(2-bromo-5-fluorophenoxy)piperidin-1-yl)isoxazol-5-yl)-2H-tetrazol-2-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-8245 50 mg (Experimental): MK-8245, 50 mg, twice daily for 28 days
  Interventions: Drug: MK-8245
- Placebo (Placebo Comparator): Placebo to MK-8245, 50 mg, twice daily
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: MK-8245 — MK-8245 50 mg twice daily for 28 days
  Arms: MK-8245 50 mg
Drug: Comparator: placebo — matching placebo to MK-8245 twice daily for 28 days
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics, and glucose lowering activity of MK-8245 in participants with type 2 diabetes. The primary hypothesis of the study is that after 4 weeks of treatment, MK-8245 produces a greater reduction in 24 hour weighted mean glucose (WMG) from baseline than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of type 2 diabetes and is being treated with diet and exercise alone, a single oral anti-hyperglycemic agent or a combination of two oral anti-hyperglycemic agents
* Subject is willing to follow a weight-maintaining diet and exercise program during the study
* Subject is a nonsmoker or is willing to limit smoking to 10 cigarettes per day while in the clinical research unit

Exclusion Criteria:

* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of cancer, except certain skin and cervical cancers or cancer that was successfully treated 10 or more years prior to screening
* Subject has a history of type 1 diabetes
* Subject has used contact lenses within the last 6 months
* Subject has used any lipid-lowering therapy in the last 3 months, except statins, Zetia, or Vytorin
* Subject has more than 3 alcoholic beverages per day
* Subject has more than 6 servings of caffeine a day
* Subject has participated in a previous MK8245 study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-08-24 (Actual); Primary Completion 2010-01-12 (Actual); Study Completion 2010-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=8245-012&kw=8245-012&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study in 5 clinical centers in the United States.
Groups:
- MK-8245 100 mg: MK-8245, 50 mg, twice daily for 28 days
- Placebo: Placebo to MK-8245, twice daily for 28 days
Period: Overall Study
Arm/Group | MK-8245 100 mg | Placebo
Started | 28 | 28
Completed | 25 | 25
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Positive drug screen | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Consistently high glucose values | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8245 100 mg | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (8.53) | 52.7 (7.30) | 53.7 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-hour Weighted Mean Glucose (WMG)
Description: The 24-hour WMG is derived from multiple glucose values collected during both fasting and post-meal periods. A "weighted" rather than a "simple" mean is used to avoid overrepresentation of post-meal glucose values. Blood samples for glucose were collected immediately prior to, and after each meal, and overnight and fasting one hour pre-dose.
Time Frame: Baseline and Day 28
Population: All participants who were compliant with the study procedures and have available data from at least one treatment were included in the primary analysis dataset.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-8245 100 mg | Placebo
Number analyzed (Participants) | 25 | 26
mg/dL | 11.0 (27.6) | -4.4 (31.7)
Statistical Analysis 1: Comparison: MK-8245 100 mg vs Placebo; Test type: Superiority or Other; p = 0.083, Least Squares Means Difference; Mean Difference (Final Values) = -15.34, 90% CI 2-sided [-29.87 to -0.82], Standard Error of Mean 8.70 — Placebo - MK-8245 on Day 28

2. Primary Outcome: Number of Participants Who Experienced Serious or Non-serious Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. A serious AE is any untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Up to Day 31
Population: All participants who received at least one dose of the investigational drug.
Measure: Number; unit: Participants
Arm/Group | MK-8245 100 mg | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  Serious Adverse Events | 0 | 0
  Non-Serious Adverse Events | 16 | 10

3. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an AE
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to Day 28
Population: All participants who received at least one dose of the investigational drug.
Measure: Number; unit: Participants
Arm/Group | MK-8245 100 mg | Placebo
Number analyzed (Participants) | 28 | 28
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to Day 31
Description: All participants who received at least one dose of the investigational drug.
Arm/Group | MK-8245 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 16/28 | 8/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-8245 100 mg (N=28) | Placebo (N=28)
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 1
Headache (Nervous system disorders) | 5 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.